CLINICAL TRIAL: NCT03441399
Title: Antidepressant Medication Adherence in Adults With Depression
Brief Title: Comparing Differing Financial Incentive Structures for Increasing Antidepressant Adherence Among Adults
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1P50MH113840-01 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Depression
Keywords: Medication Adherence
MeSH Terms: conditions — Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Escalating Incentives (Experimental): Participants assigned to the escalating financial incentives will receive an increasing financial incentive for taking their antidepressant medication for the initial 6 weeks of treatment.
  Interventions: Other: Financial incentives
- De-escalating Incentives (Experimental): Participants assigned to the de-escalating financial incentives will receive a decreasing financial incentive for taking their antidepressant medication for the initial 6 weeks of treatment.
  Interventions: Other: Financial incentives
- Control (No Intervention): Participants in this condition will receive usual care.

INTERVENTIONS:
Other: Financial incentives — Providing money for taking antidepressant medication
  Arms: De-escalating Incentives; Escalating Incentives

SUMMARY:
The investigators will test using financial incentives by leveraging decision-making biases to improve adherence to antidepressants among adults newly prescribed antidepressants. This study will compare the effects of usual care, increasing financial incentives, and decreasing financial incentives on daily antidepressant medication adherence and depression symptom control of non-elderly adults with Major Depressive Disorder.

DETAILED DESCRIPTION:
A three arm randomized controlled trial will compare interventions to promote antidepressant adherence. One hundred twenty adults with major depressive disorder (MDD) who are initiating antidepressant treatment will be randomized in equal proportion to 1) usual care, 2) usual care and an escalating daily financial incentive for 6 weeks, or 3) usual care and a de-escalating financial incentive for daily antidepressant adherence for 6 weeks. Study patients will participate in three assessments over a 12 week period as well as passive monitoring of antidepressant daily adherence through a wireless electronic pill bottle over the same 12 week period. The primary outcome will be the number of antidepressant daily doses taken during the initial six weeks of treatment. The secondary outcome will be daily adherence during the next six weeks following the discontinuation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed antidepressant
* Plan to take antidepressant as prescribed
* Working cell phone that allows texting
* Score on PHQ-9 ≥ 10

Exclusion Criteria:

* No antidepressant use in last 90 days
* Never been diagnosed with bipolar disorder, schizophrenia, or schizoaffective disorder
* Not currently pregnant or breastfeeding
* No other serious medical condition

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Antidepressant adherence | Daily for first 6 weeks of study
  The number of antidepressant daily doses taken during the initial six weeks of treatment

SECONDARY OUTCOMES:
Antidepressant adherence post-intervention | Daily between 6 and 12 weeks
  The number of antidepressant daily doses taken between 6 and 12 weeks
Depression symptoms | At baseline, 6 week follow-up, and 12 week follow-up
  Severity of depressive symptoms as assessed by the Patient Health Questionnaire (PHQ-9). The PHQ-9 measures depressive symptoms, with scores ranging from 0-27 (higher scores meaning more depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Marcus, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcus SC, Reilly ME, Zentgraf K, Volpp KG, Olfson M. Effect of Escalating and Deescalating Financial Incentives vs Usual Care to Improve Antidepressant Adherence: A Pilot Randomized Clinical Trial. JAMA Psychiatry. 2021 Feb 1;78(2):222-224. doi: 10.1001/jamapsychiatry.2020.3000. PMID 32965464
- [Derived] Beidas RS, Volpp KG, Buttenheim AN, Marcus SC, Olfson M, Pellecchia M, Stewart RE, Williams NJ, Becker-Haimes EM, Candon M, Cidav Z, Fishman J, Lieberman A, Zentgraf K, Mandell D. Transforming Mental Health Delivery Through Behavioral Economics and Implementation Science: Protocol for Three Exploratory Projects. JMIR Res Protoc. 2019 Feb 12;8(2):e12121. doi: 10.2196/12121. PMID 30747719